CLINICAL TRIAL: NCT07389226
Title: The Effect of Apple Cider Vinegar Supplementation on 24-hour Urine Chemistry in Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB25-0715
Record Dates: First submitted 2026-01-27; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Kidney Stones; Urine Specimen Collection
Keywords: urine specimen collection; kidney stones
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- kidney stone patients and healthy participants (Experimental): Each participant will be asked to complete a basic metabolic panel prior to initiating the study to ensure that no baseline metabolic derangements exist. On day 1, participants will complete a 24-hour urine collection and 48-hour food diary at home. Participants will then consume an ACV gummy containing 60 meq daily for 14 consecutive days.
  Interventions: Dietary Supplement: Apple Cider Vinegar

INTERVENTIONS:
Dietary Supplement: Apple Cider Vinegar — Goli Apple Cider Vinegar gummies

SUMMARY:
This is a single-center prospective cohort study to evaluate the effect of short-term daily apple cider vinegar (ACV) supplementation on urine chemistry.

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether a two-week course of daily ACV supplementation significantly changes an individual's urine chemistry. The investigators will study this in healthy individuals and individuals with kidney stones.

ELIGIBILITY:
Inclusion Criteria:

* Controls: Adults above the age of 18.
* Kidney stone patients: Adults above the age of 18.
* History of majority (>50%) calcium oxalate kidney stones

Exclusion Criteria:

* Anyone with a history of calcium phosphate stones (>50% calcium phosphate), uric acid stones, struvite stones, recent urinary tract instrumentation (<30 days), or recurrent urinary tract infections.
* Any individual who has had ACV outside of normal consumption in the prior month will be excluded.
* Any individual who has a history of a negative reaction (increased acid reflux, allergy) to ACV will also be excluded.
* Any individual with chronic kidney disease, underlying acid base disorder will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Measure changes in citrate in urine. | From Enrollment to 2 weeks
  to evaluate the effect of short-term daily apple cider vinegar (ACV) supplementation on urine chemistry.
Measure changes in Urine PH | From enrollment to 2 weeks
  to evaluate the effect of short-term daily apple cider vinegar (ACV) supplementation on urine chemistry.
Measure changes in calcium in urine. | from enrollment to 2 weeks
  to evaluate the effect of short-term daily apple cider vinegar (ACV) supplementation on urine chemistry.
Measure changes in calcium oxalate in urine | From Enrollment to 2 weeks
  to evaluate the effect of short-term daily apple cider vinegar (ACV) supplementation on urine chemistry.

CONTACTS AND LOCATIONS:
Overall Officials: Luke Reynolds, Principal Investigator — The University of Chicago Medical Center
Locations (1):
- The University of Chicago, Chicago, Illinois, United States